CLINICAL TRIAL: NCT05067933
Title: A Phase 2, Double-Blind, Multi-Center, Randomized, Placebo-Controlled, Dose-Ranging Trial to Determine the Safety, Immunogenicity and Efficacy of an Adenoviral-Vector Based Vaccine Expressing Severe Acute Respiratory Syndrome (SARS-CoV-2) and dsRNA Adjuvant Administered Orally
Brief Title: A Ph 2 Trial With an Oral Tableted COVID-19 Vaccine
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study drug was no longer available.
Sponsor: Vaxart (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Prevention
Other Study IDs: VXA-COV2-201
Record Dates: First submitted 2021-09-16; First posted 2021-10-05 (Actual); Results first posted 2025-04-13 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-03

CONDITIONS: COVID-19
Keywords: oral vaccine; SARS-CoV-2; tablet vaccine
MeSH Terms: conditions — COVID-19 | interventions — VXA-CoV2-1.1-S vaccine

STUDY DESIGN:
Intervention Model Description: Open-label dose and age escalation lead in phase in naive and prior vaccinated subjects, followed by a multi-center, placebo-controlled efficacy phase.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-Blind, Randomized (Part 2)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Part 1 Cohort 1a (Naïve, low dose, young adult) (Experimental): 1E10 repeat-dose vaccinations with VXA-CoV2-1.1-S at Days 1 and 29 in young adults (18-55 yrs) who are vaccine naïve
  Interventions: Drug: VXA-CoV2-1.1-S
- Part 1 Cohort 1b (Naïve, high dose, young adult) (Experimental): 1E11 repeat-dose vaccinations with VXA-CoV2-1.1-S at Days 1 and 29 in young adults (18-55 yrs) who are vaccine naïve
  Interventions: Drug: VXA-CoV2-1.1-S
- Part 1 Cohort 1c (Naïve, low dose, older adult) (Experimental): 1E10 repeat-dose vaccinations with VXA-CoV2-1.1-S at Days 1 and 29 in older adults (56-75 yrs) who are vaccine naïve
  Interventions: Drug: VXA-CoV2-1.1-S
- Part 1 Cohort 1d (Naïve, high dose, older adult) (Experimental): 1E11 repeat-dose vaccinations with VXA-CoV2-1.1-S at Days 1 and 29 in older adults (56-75 yrs) who are vaccine naïve
  Interventions: Drug: VXA-CoV2-1.1-S
- Part 1 Cohort 2a (Prior vaccinated, low dose, young adult) (Experimental): 1E10 repeat-dose vaccinations with VXA-CoV2-1.1-S at Days 1 and 29 in young adults (18-55 yrs) who have received prior vaccinations with an mRNA vaccine
  Interventions: Drug: VXA-CoV2-1.1-S
- Part 1 Cohort 2b (Prior vaccinated, high dose, young adult) (Experimental): 1E11 repeat-dose vaccinations with VXA-CoV2-1.1-S at Days 1 and 29 in young adults (18-55 yrs) who have received prior vaccinations with an mRNA vaccine
  Interventions: Drug: VXA-CoV2-1.1-S
- Part 1 Cohort 2c (Prior vaccinated, low dose, older adult) (Experimental): 1E10 repeat-dose vaccinations with VXA-CoV2-1.1-S at Days 1 and 29 in older adults (56-75 yrs) who have received prior vaccinations with an mRNA vaccine
  Interventions: Drug: VXA-CoV2-1.1-S
- Part 1 Cohort 2d (Prior vaccinated, high dose, older adult) (Experimental): 1E11 repeat-dose vaccinations with VXA-CoV2-1.1-S at Days 1 and 29 in older adults (56-75 yrs) who have received prior vaccinations with an mRNA vaccine
  Interventions: Drug: VXA-CoV2-1.1-S
- Part 2 Healthy Adults: Active vaccine (Experimental): Repeat dose vaccinations with VXA-CoV2-1.1-S at dose selected from Part 1 in healthy male and female adult volunteers 18 to 75 years old
  Interventions: Drug: VXA-CoV2-1.1-S
- Part 2 Healthy Adults: Placebo control (Placebo Comparator): Repeat dose administration with matching placebo tablets in healthy male and female adult volunteers 18 to 75 years old
  Interventions: Other: Placebo Tablets

INTERVENTIONS:
Drug: VXA-CoV2-1.1-S — COVID-19 (SARS-CoV-2) E1-/E3-Deleted Replication Defective Recombinant Adenovirus 5 with dsRNA Adjuvant Oral Tablet Vaccine
  Other Names: Oral Tableted Ad5 COVID-19 Vaccine
  Arms: Part 1 Cohort 1a (Naïve, low dose, young adult); Part 1 Cohort 1b (Naïve, high dose, young adult); Part 1 Cohort 1c (Naïve, low dose, older adult); Part 1 Cohort 1d (Naïve, high dose, older adult); Part 1 Cohort 2a (Prior vaccinated, low dose, young adult); Part 1 Cohort 2b (Prior vaccinated, high dose, young adult); Part 1 Cohort 2c (Prior vaccinated, low dose, older adult); Part 1 Cohort 2d (Prior vaccinated, high dose, older adult); Part 2 Healthy Adults: Active vaccine
Other: Placebo Tablets — Placebo tablets matching the active vaccine tablets
  Arms: Part 2 Healthy Adults: Placebo control

SUMMARY:
Part 1: An open label, dose and age escalation phase to evaluate the safety and immunogenicity of VXA-CoV2-1.1-S with a repeat-dose vaccination schedule in healthy adults aged 18 - 75 years old that are either vaccine naive or have received prior vaccination with an mRNA (messenger ribonucleic acid) vaccine for the prevention of COVID-19.

Part 2: This phase will assess the efficacy of prophylactic VXA-CoV2-1.1-S against confirmed COVID-19 occurring from 7 days after second dose with a repeat-dose vaccination schedule in healthy adults compared to placebo. Safety and immunogenicity of VXA-CoV2-1.1-S will also be evaluated in this phase.

DETAILED DESCRIPTION:
Part 1: This is an open-label, dose-ranging phase of the study to determine the safety and immunogenicity of an orally administered adenoviral-vector based vaccine (VXA-COV2-1.1-S) expressing a SARS-CoV-2 antigen and dsRNA adjuvant. Post screening activities, healthy adult volunteers, either naïve or prior vaccinated with an mRNA COVID-19 vaccine, aged 18 - 55 yrs old, and then 56 - 75 yrs old, will be enrolled into the study in 8 subgroups. Participants will receive either a low or a high dose of an oral tableted vaccine at Days 1 and Day 29. The total study period will last ~ 2 months during the active phase, with a total 12 month safety follow-up period post last vaccination. Safety, reactogenicity and immunogenicity assessments will be performed at set times during the study active and follow-up periods. Subjects will be monitored for symptoms of COVID-19 throughout the duration of the study follow-up period. An independent data monitoring committee (IDMC) will provide safety oversight through the duration of the trial. Safety and immunogenicity data will inform on the dose selection for Part 2.

Part 2: This will be a placebo-controlled phase with the vaccine dose level selected from Part 1. Subjects will receive two doses of vaccine or placebo at Days 1 and 29. Subjects will be followed as in Part 1 for safety and immunogenicity. They will also be followed for 6 months for efficacy.

ELIGIBILITY:
Inclusion Criteria

1. 18 - 75 years of age (inclusive) at the time of signing the Informed Consent Form (ICF).
2. Cohort 1 ONLY - Naive of any prior vaccination for the prevention of COVID-19 (tested using a rapid antibody test) at screening and within 7 days prior to the enrollment (Day 1).
3. Cohort 2 ONLY - Have received prior immunizations (both doses) with an EUA or FDA approved mRNA vaccine for the prevention of COVID-19, at least 6 months prior to enrollment (Day 1).
4. In stable and good health, without significant medical illness, based on medical history, physical examination, vital signs, and clinical laboratory tests as determined by the Investigator.
5. Safety laboratory values1 within the following range criteria at screening:

   1. Laboratory values within normal range or grade 1 outside the range of normal with no clinical significance (NCS) for the following analytes:, alanine aminotransferase (ALT), aspartate aminotransferase (AST), and bilirubin, blood urea nitrogen (BUN), creatinine, glucose, potassium, and sodium
   2. Laboratory values within normal range for platelet counts2 and the following coagulation tests: PT/INR, aPTT and fibrinogen
6. Body mass index (BMI) between 17 and 32 kg/m2 at screening.
7. Capable of providing signed informed consent.
8. Available for all planned visits and phone calls, and willing to complete all protocol-defined procedures and assessments (including ability and willingness to swallow multiple small enteric-coated tablets per vaccine dose).

   Gender and Reproductive Considerations
9. Male or female participants. Contraception use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies. Refer to Appendix 4 (Section 9.4).
10. Female participants must not be breastfeeding and must have a negative pregnancy test at screening and before each vaccination and fulfill one of the following criteria:

    1. At least 1 year post-menopausal (defined as amenorrhea for ≥12 consecutive months prior to Screening without an alternative medical cause).

       Women under 60 years will need to verify post-menopausal status via a follicle-stimulating hormone (FSH) test if another option to prevent potential pregnancy will not be utilized for 30 days prior to baseline vaccination and until 60 days after the last vaccination.
    2. Surgically sterile
    3. Use of oral, implantable, transdermal or injectable contraceptives for 30 days prior to initial vaccination and until 60 days after the last vaccination.
    4. A reliable form of contraception must be approved by the Investigator (e.g., double barrier method, Depo-Provera, intrauterine device, Norplant, oral contraceptives, contraceptive patches).
    5. Not be sexually active (abstinent) or be in a relationship with partner who is sterile (must be discussed with site staff and documented).

Exclusion Criteria Medical Conditions

1. Clinically significant acute illness within 72 hours prior to vaccination defined as the presence of a moderate or severe illness (as determined by the Investigator through medical history and physical exam) (assessment may be repeated during screening period).
2. Current or known previous infection with SARS-CoV-2 or receipt of any therapeutic for the prevention or treatment of COVID-19, Middle East Respiratory Syndrome (MERS), or severe acute respiratory syndrome (SARS). [EUA or FDA approved mRNA vaccines for the prevention of SARS-CoV-2 infection taken at least 6 months prior to enrollment are permitted in Cohort 2]
3. Individuals with the following underlying medical conditions who are at higher risk (or might be at higher risk) of severe illness from COVID-19 per the guidance from the Centers for Disease Control and Prevention (CDC):

   1. Cancer, including history of cancer or treatment within past 3 years (excluding basal cell carcinoma or squamous cell carcinoma)
   2. Chronic kidney disease
   3. Chronic obstructive pulmonary disease (COPD)
   4. Immunocompromised state from solid organ transplant, or other medical condition
   5. Serious heart conditions, such as heart failure, coronary artery disease, or cardiomyopathies
   6. Sickle cell disease
   7. Uncontrolled type 2 diabetes mellitus
   8. Asthma (moderate to severe)
   9. Cerebrovascular disease
   10. Cystic fibrosis
   11. Uncontrolled hypertension or high blood pressure
   12. Immunocompromised state from blood or bone marrow transplant, immune deficiencies, HIV, use of corticosteroids, or use of other immune weakening medicines
   13. Neurologic conditions, such as dementia
   14. Liver disease
   15. Pregnancy or breast feeding
   16. Pulmonary fibrosis
   17. Chronic smoking (≥ 1 cigarette per day)
   18. Thalassemia
   19. Type 1 diabetes mellitus
4. Diagnosed bleeding disorder or significant bruising or bleeding difficulties that could make blood draws problematic.
5. Any condition that resulted in the absence or removal of the spleen.
6. Any other condition that in the clinical judgment of the Investigator would jeopardize the safety or rights of a participant participating in the study, would render the participant unable to comply with the protocol or would interfere with the evaluation of the study endpoints.

   Diagnostic Assessments
7. Temperature ≥38.0ºC (100.4°F) within 24 hours prior to the planned study vaccination (assessment may be repeated during screening period).
8. Positive HIV, Hepatitis B surface antigen (HBsAg) or HCV tests at the screening visit.
9. History of gastrointestinal bleeding (e.g. melena or hematochezia) Prior/Concurrent Therapy Note: The Active Period is defined as the time period from Day 1 through Week 8, or 4 weeks post last vaccination.
10. Receipt of a licensed influenza vaccine within 14 days prior to baseline vaccination or another licensed vaccine within 28 days prior to baseline vaccination, or planned administration during the study active period.
11. Use of antiviral medications , including anti-retrovirals within 1 week before vaccination or planned use during the active study period.
12. Use of antibiotics, proton pump inhibitors, H2 blockers or antacids within 1 week before vaccination or planned use during the active study period.
13. Use of medications known to affect the immune function (e.g., systemic corticosteroids and others) within 14 days before vaccination or planned use during the active study period.
14. Daily use of nonsteroidal anti-inflammatory drugs, sulfonylureas, and angiotensin II blockers within 1 week before vaccination or planned use during the active study period.
15. Positive urine drug screen for drugs of abuse at screening (except for previous marijuana use); concurrent or planned use of marijuana during the active study period.
16. Administration of any investigational vaccine, drug or device within 8 weeks preceding vaccination, or planned use within the duration of the study.

    Other Exclusions
17. Donation or use of blood or blood products within 4 weeks prior to vaccination or planned donation during the study period.
18. Any significant hospitalization within the last year which in the opinion of the Investigator or Sponsor could interfere with study participation.
19. History of drug, alcohol or chemical abuse within 1 year of screening.
20. History of hypersensitivity or allergic reaction to any component of the investigational vaccine, including but not limited to fish gelatin.
21. Any of the following history or conditions that may lead to higher risk of clotting events and/or thrombocytopenia:

    1. Family or personal history of bleeding or thrombosis
    2. History of heparin-related thrombotic events, and/or receiving heparin treatments
    3. History of autoimmune or inflammatory disease
    4. Presence of any of the following conditions known to increase risk of thrombosis within 6 months prior to screening:

       * Recent surgery other than removal/biopsy of cutaneous lesions
       * Immobility (confined to bed or wheelchair for 3 or more successive days)
       * Head trauma with loss of consciousness or documented brain injury
       * Receipt of anticoagulants for prophylaxis of thrombosis
       * Recent clinically significant infection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2021-10-22 (Actual); Primary Completion 2022-06-10 (Actual); Study Completion 2023-05-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Cummings, MD, Study Director — Vaxart, Inc.
Locations (4):
- United States (4):
  - Ark Clinical Research, Long Beach, California
  - AMR Wichita East, Wichita, Kansas
  - Velocity Clinical Research, Inc,, Cleveland, Ohio
  - AMR Knoxville, Knoxville, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 66 participants were enrolled at 5 sites in the United States between 22 October 2021 and 09 May 2023 (follow-up period cut-off) in Part 1 of the study.
  Vaxart decided not to conduct Part 2 of this study, so results for Part 2 were not included in this summary.
Groups:
- Cohort 1a: Vaccine Naïve, 18-55 Years, Low-dose: Healthy, vaccine naïve participants aged between 18 and 55 years received VXA-CoV2-1.1-S at a dose of 1 x 10^10 infectious units (IU) ± 0.5 log as an oral tablet on Day 1 and Day 29 of the 57-day active study period. Participants then entered the safety follow-up period until Month 13.
- Cohort 1b: Vaccine Naïve, 18-55 Years, High-dose: Healthy, vaccine naïve participants aged between 18 and 55 years received VXA-CoV2-1.1-S at a dose of 1 x 10^11 IU ± 0.5 log as an oral tablet on Day 1 and Day 29 of the 57-day active study period. Participants then entered the safety follow-up period until Month 13.
- Cohort 1c: Vaccine Naïve, 56-75 Years, Low-dose: Healthy, vaccine naïve participants aged between 56 and 75 years received VXA-CoV2-1.1-S at a dose of 1 x 10^10 IU ± 0.5 log as an oral tablet on Day 1 and Day 29 of the 57-day active study period. Participants then entered the safety follow-up period until Month 13.
- Cohort 2a: Prior Vaccinated, 18-55 Years, Low-dose: Healthy, prior vaccinated participants aged between 18 and 55 years received VXA-CoV2-1.1-S at a dose of 1 x 10^10 IU ± 0.5 log as an oral tablet on Day 1 and Day 29 of the 57-day active study period. Participants then entered the safety follow-up period until Month 13.
- Cohort 2b: Prior Vaccinated, 18-55 Years, High-dose: Healthy, prior vaccinated participants aged between 18 and 55 years received VXA-CoV2-1.1-S at a dose of 1 x 10^11 IU ± 0.5 log as an oral tablet on Day 1 and Day 29 of the 57-day active study period. Participants then entered the safety follow-up period until Month 13.
- Cohort 2c: Prior Vaccinated, 56-75 Years, Low-dose: Healthy, prior vaccinated participants aged between 56 and 75 years received VXA-CoV2-1.1-S at a dose of 1 x 10^10 IU ± 0.5 log as an oral tablet on Day 1 and Day 29 of the 57-day active study period. Participants then entered the safety follow-up period until Month 13.
Period: Overall Study
Arm/Group | Cohort 1a: Vaccine Naïve, 18-55 Years, Low-dose | Cohort 1b: Vaccine Naïve, 18-55 Years, High-dose | Cohort 1c: Vaccine Naïve, 56-75 Years, Low-dose | Cohort 2a: Prior Vaccinated, 18-55 Years, Low-dose | Cohort 2b: Prior Vaccinated, 18-55 Years, High-dose | Cohort 2c: Prior Vaccinated, 56-75 Years, Low-dose
Started | 12 | 9 | 8 | 13 | 12 | 12
Received First Dose of VXA-CoV2-1.1-S | 12 | 9 | 8 | 13 | 12 | 12
Received Both Doses of VXA-CoV2-1.1-S | 11 | 9 | 8 | 13 | 12 | 12
Entered Safety Follow-up Period | 10 | 9 | 8 | 12 | 12 | 12
Completed | 8 | 8 | 7 | 10 | 11 | 12
Not Completed | 4 | 1 | 1 | 3 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 1 | 2 | 1 | 0
Not completed — Miscellaneous | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population: Included all randomized participants who received at least one dose of the study drug and were analyzed in the treatment group corresponding to actual study drug received. Participant flow is presented per cohort due to sequential enrollment. As pre-specified in Protocol Section 8.3, Baseline Characteristics, Outcome Measures and Adverse Event analysis were summarized by vaccine group according to the study drugs they actually received.
Groups:
- VXA-CoV2-1.1-S: 1 x 10^10 IU ± 0.5 Log: Healthy participants received VXA-CoV2-1.1-S at a dose of 1 x 10^10 IU ± 0.5 log as an oral tablet on Day 1 and Day 29 of the 57-day active study period. Participants then entered the safety follow-up period until Month 13.
- VXA-CoV2-1.1-S: 1 x 10^11 IU ± 0.5 Log: Healthy participants received VXA-CoV2-1.1-S at a dose of 1 x 10^11 IU ± 0.5 log as an oral tablet on Day 1 and Day 29 of the 57-day active study period. Participants then entered the safety follow-up period until Month 13.
- Total: Total of all reporting groups
Arm/Group | VXA-CoV2-1.1-S: 1 x 10^10 IU ± 0.5 Log | VXA-CoV2-1.1-S: 1 x 10^11 IU ± 0.5 Log | Total
Number analyzed (Participants) | 45 | 21 | 66
Age, Customized [Count of Participants; unit: Participants]
  18 - 55 years | 25 | 21 | 46
  56 - 75 years | 20 | 0 | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 10 | 30
  Male | 25 | 11 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 5 | 15
  Not Hispanic or Latino | 35 | 16 | 51
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 29 | 10 | 39
  Black or African American | 6 | 5 | 11
  Asian | 6 | 4 | 10
  Other | 2 | 1 | 3
  Multiple | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced a Solicited Symptom of Reactogenicity
Description: Solicited symptoms of reactogenicity were predefined systemic signs and symptoms of reactogenicity for which the participant was specifically questioned, and which were noted by the participant in their daily Solicited Symptom Diary for 7 days after each vaccination, including:
  * fever (any temperature 100°F or higher)
  * headache
  * myalgia (muscle pain)
  * abdominal pain
  * anorexia (defined and not eating)
  * nausea
  * vomiting
  * diarrhea
  * malaise/fatigue
Time Frame: Up to 7 days after Dose 1 (Days 1 to 8) and Dose 2 (Days 29 to 36)
Population: Safety Population: Included all randomized participants who received at least one dose of the study drug. Only participants with evaluable data at each dosing time point were included. As pre-specified in Protocol Section 8.3, Baseline Characteristics, Outcome Measures and Adverse Event analysis were summarized by vaccine group according to the study drugs they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | VXA-CoV2-1.1-S: 1 x 10^10 IU ± 0.5 Log | VXA-CoV2-1.1-S: 1 x 10^11 IU ± 0.5 Log
Number analyzed (Participants) | 45 | 21
Participants
  Dose 1 | 16 | 10
  Dose 2: number analyzed (Participants) | 44 | 21
  Dose 2 | 13 | 4

2. Primary Outcome: Severity of Solicited Symptoms of Reactogenicity
Description: Solicited symptoms of reactogenicity were predefined systemic signs and symptoms of reactogenicity for which the participant was specifically questioned, and which were noted by the participant in their daily Solicited Symptom Diary for 7 days after each vaccination, including:
  * fever (any temperature 100°F or higher)
  * headache
  * myalgia (muscle pain)
  * abdominal pain
  * anorexia (defined and not eating)
  * nausea
  * vomiting
  * diarrhea
  * malaise/fatigue
  Participants were instructed to rate solicited symptoms of reactogenicity that were collected in their Solicited Symptom Diary with the below grades, against pre-defined criteria as noted in the protocol:
  * Grade 1 - Mild
  * Grade 2 - Moderate
  * Grade 3 - Severe
  * Grade 4 - Life Threatening
  Participants with multiple solicited symptoms were only counted once, the highest severity of which was used.
Time Frame: Up to 7 days after Dose 1 (Days 1 to 8) and Dose 2 (Days 29 to 36)
Population: Safety Population: Included all randomized participants who received at least one dose of the study drug and experienced a solicited symptom of reactogenicity. As pre-specified in Protocol Section 8.3, Baseline Characteristics, Outcome Measures and Adverse Event analysis were summarized by vaccine group according to the study drugs they actually received. The overall number of participants analyzed is inclusive of participants all participants with symptoms following Dose 1 and/or Dose 2.
Measure: Count of Participants; unit: Participants
Arm/Group | VXA-CoV2-1.1-S: 1 x 10^10 IU ± 0.5 Log | VXA-CoV2-1.1-S: 1 x 10^11 IU ± 0.5 Log
Number analyzed (Participants) | 23 | 11
Participants
  Dose 1: number analyzed (Participants) | 16 | 10
  Dose 1: Grade 1 - Mild | 11 | 8
  Dose 1: Grade 2 - Moderate | 5 | 2
  Dose 1: Grade 3 - Severe | 0 | 0
  Dose 1: Grade 4 - Life Threatening | 0 | 0
  Dose 2: number analyzed (Participants) | 13 | 4
  Dose 2: Grade 1 - Mild | 7 | 3
  Dose 2: Grade 2 - Moderate | 6 | 1
  Dose 2: Grade 3 - Severe | 0 | 0
  Dose 2: Grade 4 - Life Threatening | 0 | 0

3. Primary Outcome: Number of Participants Who Experienced an Unsolicited Treatment-emergent Adverse Event (TEAE) During the Active Treatment Period
Description: A TEAE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention, occurring after first dose of study drug.
  A serious TEAE was any TEAE that met any of the following criteria:
  * Resulted in death.
  * Was life-threatening.
  * Required inpatient hospitalization or prolongation of existing hospitalization.
  * Resulted in persistent or significant disability/incapacity.
  * Was a congenital anomaly/birth defect.
  * Was a suspected transmission of any infectious agent via a medicinal product.
  * Was a significant medical event, as judged by the investigator.
Time Frame: Day 1 to Day 57
Population: Safety Population: Included all randomized participants who received at least one dose of the study drug. As pre-specified in Protocol Section 8.3, Baseline Characteristics, Outcome Measures and Adverse Event analysis were summarized by vaccine group according to the study drugs they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | VXA-CoV2-1.1-S: 1 x 10^10 IU ± 0.5 Log | VXA-CoV2-1.1-S: 1 x 10^11 IU ± 0.5 Log
Number analyzed (Participants) | 45 | 21
Participants
  Any TEAE | 10 | 4
  Any Serious TEAE | 1 | 0

4. Primary Outcome: Severity of Unsolicited TEAEs During the Active Treatment Period
Description: All unsolicited TEAEs during the active treatment period were assessed by the investigator using the below scale:
  * Mild: Events that required minimal or no treatment and did not interfere with the participant's daily activities.
  * Moderate: Events that resulted in a low level of inconvenience or concern with the therapeutic measures. Moderate events may have caused some interference with functioning.
  * Severe: Events that interrupted a participant's usual daily activity and may have required systemic drug therapy or other treatment. Severe events were usually incapacitating.
  * Life Threatening: Any adverse drug experience that placed the participant, in the view of the investigator, at immediate risk of death from the reaction as it occurred.
  Participants with multiple TEAEs during the active treatment period were only counted once, the highest severity of which was used.
Time Frame: Day 1 to Day 57
Population: Safety Population: Included all randomized participants who received at least 1 dose of study drug & experienced an unsolicited TEAE during the active treatment period. As pre-specified in Protocol Section 8.3, Baseline Characteristics, Outcome Measures & Adverse Event analysis were summarized by vaccine group according to the study drugs they actually received. The overall number of participants analyzed is inclusive of participants all participants with symptoms following Dose 1 &/or Dose 2.
Measure: Count of Participants; unit: Participants
Arm/Group | VXA-CoV2-1.1-S: 1 x 10^10 IU ± 0.5 Log | VXA-CoV2-1.1-S: 1 x 10^11 IU ± 0.5 Log
Number analyzed (Participants) | 10 | 4
Participants
  Any TEAE: Mild | 4 | 3
  Any TEAE: Moderate | 4 | 1
  Any TEAE: Severe | 2 | 0
  Any TEAE: Life Threatening | 0 | 0
  Any Serious TEAE: number analyzed (Participants) | 1 | 0
  Any Serious TEAE: Mild | 0 | 0
  Any Serious TEAE: Moderate | 0 | 0
  Any Serious TEAE: Severe | 1 | 0
  Any Serious TEAE: Life Threatening | 0 | 0

5. Primary Outcome: Number of Participants Who Experienced a Medically Attended Adverse Event (MAAE) During the Active Treatment Period
Description: MAAEs were defined as TEAEs with medically-attended visits including hospital, emergency room, urgent care clinic, or other visits to or from medical personnel for any reason. Routine study visits were not considered medically-attended visits. New onset of chronic illness/diseases (NOCI) and adverse events of special interest (AESIs) were collected as part of the MAAEs. As defined in the protocol, adverse events for potential immune-mediated medical conditions as well as events associated with thrombosis and thrombocytopenia were considered AESIs.
Time Frame: Day 1 to Day 57
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | VXA-CoV2-1.1-S: 1 x 10^10 IU ± 0.5 Log | VXA-CoV2-1.1-S: 1 x 10^11 IU ± 0.5 Log
Number analyzed (Participants) | 45 | 21
Participants | 6 | 0

6. Primary Outcome: Severity of MAAEs During the Active Treatment Period
Description: All MAAEs during the active treatment period were assessed by the investigator using the below scale:
  * Mild: Events that required minimal or no treatment and did not interfere with the participant's daily activities.
  * Moderate: Events that resulted in a low level of inconvenience or concern with the therapeutic measures. Moderate events may have caused some interference with functioning.
  * Severe: Events that interrupted a participant's usual daily activity and may have required systemic drug therapy or other treatment. Severe events were usually incapacitating.
  * Life Threatening: Any adverse drug experience that placed the participant, in the view of the investigator, at immediate risk of death from the reaction as it occurred.
  Participants with multiple MAAEs during the active treatment period were only counted once, the highest severity of which was used.
Time Frame: Day 1 to Day 57
Population: Safety Population: Included all randomized participants who received at least one dose of the study drug. Only participants who experienced an MAAE during the active treatment period were included. As pre-specified in Protocol Section 8.3, Baseline Characteristics, Outcome Measures and Adverse Event analysis were summarized by vaccine group according to the study drugs they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | VXA-CoV2-1.1-S: 1 x 10^10 IU ± 0.5 Log | VXA-CoV2-1.1-S: 1 x 10^11 IU ± 0.5 Log
Number analyzed (Participants) | 6 | 0
Participants
  Mild | 2 |
  Moderate | 2 |
  Severe | 2 |
  Life Threatening | 0 |

7. Secondary Outcome: Number of Participants Who Experienced a MAAE During the Safety Follow-up Period
Description: MAAEs were defined as TEAEs with medically-attended visits including hospital, emergency room, urgent care clinic, or other visits to or from medical personnel for any reason. Routine study visits were not considered medically-attended visits. NOCI and AESIs were collected as part of the MAAEs. As defined in the protocol, adverse events for potential immune-mediated medical conditions as well as events associated with thrombosis and thrombocytopenia were considered AESIs.
Time Frame: From last dose up to 12 months post-last dose
Population: Safety Population: Included all randomized participants who received at least one dose of the study drug. Only participants who entered the safety follow-up period were included. As pre-specified in Protocol Section 8.3, Baseline Characteristics, Outcome Measures and Adverse Event analysis were summarized by vaccine group according to the study drugs they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | VXA-CoV2-1.1-S: 1 x 10^10 IU ± 0.5 Log | VXA-CoV2-1.1-S: 1 x 10^11 IU ± 0.5 Log
Number analyzed (Participants) | 44 | 21
Participants | 5 | 2

8. Secondary Outcome: Severity of MAAEs During the Safety Follow-up Period
Description: All MAAEs during the safety follow-up period were assessed by the investigator using the below scale:
  * Mild: Events that required minimal or no treatment and did not interfere with the participant's daily activities.
  * Moderate: Events that resulted in a low level of inconvenience or concern with the therapeutic measures. Moderate events may have caused some interference with functioning.
  * Severe: Events that interrupted a participant's usual daily activity and may have required systemic drug therapy or other treatment. Severe events were usually incapacitating.
  * Life Threatening: Any adverse drug experience that placed the participant, in the view of the investigator, at immediate risk of death from the reaction as it occurred.
  Participants with multiple MAAEs during the safety follow-up period were only counted once, the highest severity of which was used.
Time Frame: From last dose up to 12 months post-last dose
Population: Safety Population: Included all randomized participants who received at least one dose of the study drug. Only participants who experienced an MAAE during the safety follow-up period were included. As pre-specified in Protocol Section 8.3, Baseline Characteristics, Outcome Measures and Adverse Event analysis were summarized by vaccine group according to the study drugs they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | VXA-CoV2-1.1-S: 1 x 10^10 IU ± 0.5 Log | VXA-CoV2-1.1-S: 1 x 10^11 IU ± 0.5 Log
Number analyzed (Participants) | 5 | 2
Participants
  Mild | 1 | 0
  Moderate | 2 | 2
  Severe | 2 | 0
  Life Threatening | 0 | 0

9. Secondary Outcome: Number of Participants Who Experienced a Serious TEAE During the Safety Follow-up Period
Description: as for outcome 3
Time Frame: From last dose up to 12 months post-last dose
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | VXA-CoV2-1.1-S: 1 x 10^10 IU ± 0.5 Log | VXA-CoV2-1.1-S: 1 x 10^11 IU ± 0.5 Log
Number analyzed (Participants) | 44 | 21
Participants | 3 | 0

10. Secondary Outcome: Severity of Serious TEAEs During the Safety Follow-up Period
Description: All serious TEAEs during the active treatment period were assessed by the investigator using the below scale:
  * Mild: Events that required minimal or no treatment and did not interfere with the participant's daily activities.
  * Moderate: Events that resulted in a low level of inconvenience or concern with the therapeutic measures. Moderate events may have caused some interference with functioning.
  * Severe: Events that interrupted a participant's usual daily activity and may have required systemic drug therapy or other treatment. Severe events were usually incapacitating.
  * Life Threatening: Any adverse drug experience that placed the participant, in the view of the investigator, at immediate risk of death from the reaction as it occurred.
  Participants with multiple serious TEAEs during the active treatment period were only counted once, the highest severity of which was used.
Time Frame: From last-dose up to 12 months post-last dose
Population: Safety Population: Included all randomized participants who received at least one dose of the study drug. Only participants who experienced a serious TEAE during the safety follow-up period were included. As pre-specified in Protocol Section 8.3, Baseline Characteristics, Outcome Measures and Adverse Event analysis were summarized by vaccine group according to the study drugs they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | VXA-CoV2-1.1-S: 1 x 10^10 IU ± 0.5 Log | VXA-CoV2-1.1-S: 1 x 10^11 IU ± 0.5 Log
Number analyzed (Participants) | 3 | 0
Participants
  Mild | 0 |
  Moderate | 0 |
  Severe | 2 |
  Life Threatening | 1 |

11. Secondary Outcome: Levels of SARS-CoV2-specific Immunoglobulin G Spike (IgG-S) Antibodies by Mesoscale Discovery (MSD) Assay
Description: SARS-CoV2-specific IgG-S antibody levels were measured on specific timepoints via MSD assay. For results below the lower limit of quantification (LLOQ), the value was replaced with 1/2 the numeric portion of the original result rounded up to nearest integer. For results above the upper limit of quantification (ULOQ), the value was replaced with the numeric portion of the original result.
Time Frame: Day 1, Day 29 and Day 57
Population: Per Protocol Population: Included all participants who were enrolled and received at least 1 dose of study drug who were free from major protocol violations. As pre-specified in Protocol Section 8.3, Baseline Characteristics, Outcome Measures and Adverse Event analysis were summarized by vaccine group according to the study drugs they actually received.
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Arm/Group | VXA-CoV2-1.1-S: 1 x 10^10 IU ± 0.5 Log | VXA-CoV2-1.1-S: 1 x 10^11 IU ± 0.5 Log
Number analyzed (Participants) | 38 | 19
AU/mL
  Day 1 | 4708.7 [1555.28 to 14255.88] | 6323.8 [1721.12 to 23235.26]
  Day 29 | 6693.2 [2379.57 to 18826.24] | 10097.1 [2880.93 to 35388.51]
  Day 57 | 12348.6 [4974.39 to 30654.39] | 12868.1 [4124.72 to 40145.35]
Statistical Analysis 1: Comparison: VXA-CoV2-1.1-S: 1 x 10^10 IU ± 0.5 Log vs VXA-CoV2-1.1-S: 1 x 10^11 IU ± 0.5 Log; Test type: Other — Comparison between immunogenicity assay results between treatment groups on Day 57; p = 0.953, Wilcoxon rank sum tests

12. Secondary Outcome: Levels of SARS-CoV2-specific Immunoglobulin G Nucleocapsid (IgG-N) Antibodies by MSD Assay
Description: SARS-CoV2-specific IgG-N antibody levels were measured on specific timepoints via MSD assay. For results below the LLOQ, the value was replaced with 1/2 the numeric portion of the original result rounded up to nearest integer. For results above the ULOQ, the value was replaced with the numeric portion of the original result.
Time Frame: Day 1, Day 29 and Day 57
Population: Per Protocol Population: Included all participants with evaluable data at each time point who were enrolled and received at least 1 dose of study drug who were free from major protocol violations. As pre-specified in Protocol Section 8.3, Baseline Characteristics, Outcome Measures and Adverse Event analysis were summarized by vaccine group according to the study drugs they actually received.
Measure: Geometric Mean (95% Confidence Interval); unit: arbitrary units per milliliter (AU/mL)
Arm/Group | VXA-CoV2-1.1-S: 1 x 10^10 IU ± 0.5 Log | VXA-CoV2-1.1-S: 1 x 10^11 IU ± 0.5 Log
Number analyzed (Participants) | 38 | 19
arbitrary units per milliliter (AU/mL)
  Day 1 | 360.3 [189.03 to 686.76] | 1516 [560.05 to 4105.41]
  Day 29 | 593.3 [258.49 to 1361.80] | 1301.6 [511.21 to 3314.18]
  Day 57: number analyzed (Participants) | 37 | 19
  Day 57 | 898.2 [376.83 to 2140.91] | 1192.4 [504.15 to 2820.21]
Statistical Analysis 1: Comparison: VXA-CoV2-1.1-S: 1 x 10^10 IU ± 0.5 Log vs VXA-CoV2-1.1-S: 1 x 10^11 IU ± 0.5 Log; Test type: Other — Comparison between immunogenicity assay results between treatment groups on Day 57; p = 0.500, Wilcoxon rank sum tests

13. Secondary Outcome: Levels of SARS-CoV2-specific Immunoglobulin G Receptor-binding Domain (IgG-RBD) Antibodies by MSD Assay
Description: SARS-CoV2-specific IgG-RBD antibody levels were measured on specific timepoints via MSD assay. For results below the LLOQ, the value was replaced with 1/2 the numeric portion of the original result rounded up to nearest integer. For results above the ULOQ, the value was replaced with the numeric portion of the original result.
Time Frame: Day 1, Day 29 and Day 57
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Arm/Group | VXA-CoV2-1.1-S: 1 x 10^10 IU ± 0.5 Log | VXA-CoV2-1.1-S: 1 x 10^11 IU ± 0.5 Log
Number analyzed (Participants) | 38 | 19
AU/mL
  Day 1 | 2597.0 [869.40 to 7757.64] | 2570.5 [620.23 to 10653.33]
  Day 29 | 3513.2 [1228.26 to 10048.92] | 4520.7 [1133.60 to 18028.41]
  Day 57 | 6553.4 [2566.79 to 16731.71] | 5825.8 [1580.33 to 21476.45]
Statistical Analysis 1: Comparison: VXA-CoV2-1.1-S: 1 x 10^10 IU ± 0.5 Log vs VXA-CoV2-1.1-S: 1 x 10^11 IU ± 0.5 Log; Test type: Other — Comparison between immunogenicity assay results between treatment groups on Day 57; p = 0.912, Wilcoxon rank sum tests

14. Secondary Outcome: Levels of SARS-CoV2-specific Immunoglobulin A Spike (IgA-S) Antibodies by MSD Assay
Description: SARS-CoV2-specific IgA-S antibody levels were measured on specific timepoints via MSD assay. For results below the LLOQ, the value was replaced with 1/2 the numeric portion of the original result rounded up to nearest integer. For results above the ULOQ, the value was replaced with the numeric portion of the original result.
Time Frame: Day 1, Day 29 and Day 57
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Arm/Group | VXA-CoV2-1.1-S: 1 x 10^10 IU ± 0.5 Log | VXA-CoV2-1.1-S: 1 x 10^11 IU ± 0.5 Log
Number analyzed (Participants) | 38 | 19
AU/mL
  Day 1 | 928.4 [471.44 to 1828.24] | 809.8 [279.42 to 2346.95]
  Day 29 | 1184.5 [591.59 to 2371.69] | 1252.3 [439.64 to 3567.14]
  Day 57 | 1595.4 [812.45 to 3132.98] | 1302.9 [495.27 to 3427.63]
Statistical Analysis 1: Comparison: VXA-CoV2-1.1-S: 1 x 10^10 IU ± 0.5 Log vs VXA-CoV2-1.1-S: 1 x 10^11 IU ± 0.5 Log; Test type: Other — Comparison between immunogenicity assay results between treatment groups on Day 57; p = 0.678, Wilcoxon rank sum tests

15. Secondary Outcome: Levels of SARS-CoV2-specific Immunoglobulin A Nucleocapsid (IgA-N) Antibodies by MSD Assay
Description: SARS-CoV2-specific IgA-N antibody levels were measured on specific timepoints via MSD assay. For results below the LLOQ, the value was replaced with 1/2 the numeric portion of the original result rounded up to nearest integer. For results above the ULOQ, the value was replaced with the numeric portion of the original result.
Time Frame: Day 1, Day 29 and Day 57
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Arm/Group | VXA-CoV2-1.1-S: 1 x 10^10 IU ± 0.5 Log | VXA-CoV2-1.1-S: 1 x 10^11 IU ± 0.5 Log
Number analyzed (Participants) | 38 | 19
AU/mL
  Day 1 | 355.2 [231.48 to 544.98] | 312.9 [163.61 to 598.51]
  Day 29: number analyzed (Participants) | 37 | 19
  Day 29 | 367.8 [234.69 to 576.46] | 264.9 [135.00 to 519.69]
  Day 57 | 449.0 [275.63 to 731.52] | 260.5 [135.01 to 502.78]
Statistical Analysis 1: Comparison: VXA-CoV2-1.1-S: 1 x 10^10 IU ± 0.5 Log vs VXA-CoV2-1.1-S: 1 x 10^11 IU ± 0.5 Log; Test type: Other — Comparison between immunogenicity assay results between treatment groups on Day 57; p = 0.257, Wilcoxon rank sum tests

16. Secondary Outcome: Levels of SARS-CoV2-specific Immunoglobulin A Receptor-binding Domain (IgA-RBD) Antibodies by MSD Assay
Description: SARS-CoV2-specific IgA-RBD antibody levels were measured on specific timepoints via MSD assay. For results below the LLOQ, the value was replaced with 1/2 the numeric portion of the original result rounded up to nearest integer. For results above the ULOQ, the value was replaced with the numeric portion of the original result.
Time Frame: Day 1, Day 29 and Day 57
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Groups:
- VXA-CoV2-1.1-S: 1 x 10^11 IU ± 0.5 Log: Healthy participants received a high dose of VXA-CoV2-1.1-S at a dose of 1 x 10^11 IU ± 0.5 log as an oral tablet on Day 1 and Day 29 of the 57-day active study period. Participants then entered the safety follow-up period until Month 13.
Arm/Group | VXA-CoV2-1.1-S: 1 x 10^10 IU ± 0.5 Log | VXA-CoV2-1.1-S: 1 x 10^11 IU ± 0.5 Log
Number analyzed (Participants) | 38 | 19
AU/mL
  Day 1 | 745.1 [419.15 to 1324.62] | 562.7 [226.59 to 1397.27]
  Day 29 | 893.5 [486.55 to 1640.83] | 913.9 [378.36 to 2207.31]
  Day 57 | 1122.2 [620.31 to 2030.32] | 875.9 [379.89 to 2019.74]
Statistical Analysis 1: Comparison: VXA-CoV2-1.1-S: 1 x 10^10 IU ± 0.5 Log vs VXA-CoV2-1.1-S: 1 x 10^11 IU ± 0.5 Log; Test type: Other — Comparison between immunogenicity assay results between treatment groups on Day 57; p = 0.748, Wilcoxon rank sum tests

17. Secondary Outcome: Levels of Neutralizing Serum Antibody Titers to SARS-CoV-2
Description: Neutralizing Serum Antibody Titers to SARS-CoV-2 were measured on specific timepoints via qualified pseudovirus assay. For results below the LLOQ, the value was replaced with 1/2 the numeric portion of the original result rounded up to nearest integer. For results above the ULOQ, the value was replaced with the numeric portion of the original result.
Time Frame: Day 1, Day 29 and Day 57
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Arm/Group | VXA-CoV2-1.1-S: 1 x 10^10 IU ± 0.5 Log | VXA-CoV2-1.1-S: 1 x 10^11 IU ± 0.5 Log
Number analyzed (Participants) | 38 | 19
AU/mL
  Day 1 | 101.2 [44.16 to 231.70] | 81.7 [23.85 to 279.97]
  Day 29 | 123.6 [53.91 to 283.52] | 129.5 [39.56 to 423.61]
  Day 57 | 150.2 [62.45 to 361.09] | 147.2 [43.36 to 499.71]
Statistical Analysis 1: Comparison: VXA-CoV2-1.1-S: 1 x 10^10 IU ± 0.5 Log vs VXA-CoV2-1.1-S: 1 x 10^11 IU ± 0.5 Log; Test type: Other — Comparison between immunogenicity assay results between treatment groups on Day 57; p = 0.946, Wilcoxon rank sum tests

18. Secondary Outcome: Mean Percentage of Cluster of Differentiation 8 (CD8) T-cells Making Tumor Necrosis Factor (TNF) Alpha+ Spike (S) as Measured by Intracellular Cytokine Cytometry (ICC)
Description: Mean Percentage of CD8 T-cells making TNF alpha+S were measured on specific timepoints via ICC. For results below the LLOQ, the value was replaced with 1/2 the numeric portion of the original result rounded up to nearest integer. For results above the ULOQ, the value was replaced with the numeric portion of the original result.
Time Frame: Day 1, Day 8, Day 29 and Day 36
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: percentage of CD8 T-cells
Arm/Group | VXA-CoV2-1.1-S: 1 x 10^10 IU ± 0.5 Log | VXA-CoV2-1.1-S: 1 x 10^11 IU ± 0.5 Log
Number analyzed (Participants) | 30 | 15
percentage of CD8 T-cells
  Day 1 | 0.071 (0.1352) | 0.081 (0.0999)
  Day 8 | 0.046 (0.0750) | 0.009 (0.0234)
  Day 29: number analyzed (Participants) | 28 | 15
  Day 29 | 0.080 (0.1671) | 0.089 (0.1538)
  Day 36: number analyzed (Participants) | 21 | 10
  Day 36 | 0.067 (0.0702) | 0.122 (0.2132)

19. Secondary Outcome: Mean Percentage of CD8 T-cells Making Interferon (IFN) Gamma+S as Measured by ICC
Description: Mean Percentage of CD8 T-cells making IFN gamma+S were measured on specific timepoints via ICC. For results below the LLOQ, the value was replaced with 1/2 the numeric portion of the original result rounded up to nearest integer. For results above the ULOQ, the value was replaced with the numeric portion of the original result.
Time Frame: Day 1, Day 8, Day 29 and Day 36
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: percentage of CD8 T-cells
Arm/Group | VXA-CoV2-1.1-S: 1 x 10^10 IU ± 0.5 Log | VXA-CoV2-1.1-S: 1 x 10^11 IU ± 0.5 Log
Number analyzed (Participants) | 30 | 15
percentage of CD8 T-cells
  Day 1 | 0.349 (0.2933) | 0.440 (0.4038)
  Day 8 | 0.287 (0.3369) | 0.308 (0.4340)
  Day 29: number analyzed (Participants) | 28 | 15
  Day 29 | 0.517 (0.5043) | 0.536 (0.5142)
  Day 36: number analyzed (Participants) | 21 | 10
  Day 36 | 0.712 (0.6597) | 0.608 (0.5592)

20. Secondary Outcome: Levels of SARS-CoV2-specific IgA-S Antibodies in Nasal Swabs
Description: SARS-CoV2-specific IgA-S antibody levels in nasal swabs were measured on specific timepoints via MSD assay. For results below the LLOQ, the value was replaced with 1/2 the numeric portion of the original result rounded up to nearest integer. For results above the ULOQ, the value was replaced with the numeric portion of the original result.
Time Frame: Day 1, Day 29 and Day 57
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: AU IgA/ng Total IgA
Arm/Group | VXA-CoV2-1.1-S: 1 x 10^10 IU ± 0.5 Log | VXA-CoV2-1.1-S: 1 x 10^11 IU ± 0.5 Log
Number analyzed (Participants) | 38 | 19
AU IgA/ng Total IgA
  Day 1 | 0.142 (0.3723) | 0.102 (0.1648)
  Day 29: number analyzed (Participants) | 37 | 18
  Day 29 | 0.874 (2.9889) | 0.091 (0.1178)
  Day 57 | 0.203 (0.5061) | 0.374 (1.4455)
Statistical Analysis 1: Comparison: VXA-CoV2-1.1-S: 1 x 10^10 IU ± 0.5 Log vs VXA-CoV2-1.1-S: 1 x 10^11 IU ± 0.5 Log; Test type: Other — Comparison between immunogenicity assay results between treatment groups on Day 57; p = 0.356, Wilcoxon rank sum tests

21. Secondary Outcome: Levels of SARS-CoV2-specific IgA-S Antibodies in Saliva Swabs
Description: SARS-CoV2-specific IgA-S antibody levels in saliva swabs were measured on specific timepoints via MSD assay. For results below the LLOQ, the value was replaced with 1/2 the numeric portion of the original result rounded up to nearest integer. For results above the ULOQ, the value was replaced with the numeric portion of the original result.
Time Frame: Day 1, Day 29 and Day 57
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: AU IgA/ng Total IgA
Groups:
- VXA-CoV2-1.1-S: 1 x 10^10 IU ± 0.5 Log: Healthy participants received VXA-CoV2-1.1-S at a dose of 1 x 10^11 IU ± 0.5 log as an oral tablet on Day 1 and Day 29 of the 57-day active study period. Participants then entered the safety follow-up period until Month 13.
- VXA-CoV2-1.1-S: High Dose: Healthy participants received a high dose of VXA-CoV2-1.1-S as an oral tablet on Day 1 and Day 29 of the 57-day active study period. Participants then entered the safety follow-up period until Month 13.
Arm/Group | VXA-CoV2-1.1-S: 1 x 10^10 IU ± 0.5 Log | VXA-CoV2-1.1-S: High Dose
Number analyzed (Participants) | 38 | 19
AU IgA/ng Total IgA
  Day 1 | 0.028 (0.0341) | 0.062 (0.1541)
  Day 29 | 0.070 (0.2479) | 0.048 (0.0883)
  Day 57 | 0.058 (0.1275) | 0.047 (0.0652)
Statistical Analysis 1: Comparison: VXA-CoV2-1.1-S: 1 x 10^10 IU ± 0.5 Log vs VXA-CoV2-1.1-S: High Dose; Test type: Other — Comparison between immunogenicity assay results between treatment groups on Day 57; p = 0.267, Wilcoxon rank sum tests

ADVERSE EVENTS:
Time Frame: Active Study Period: Day 1 to Day 57; Safety Follow-up Period: Last-dose to up to 12 months post-last dose
Description: Safety Population: Included all randomized participants who received at least one dose of the study drug and were analyzed in the treatment group corresponding to actual study drug received. During the safety follow-up period, only SAEs and MAAEs were collected.
Groups:
- Active Study Period: VXA-CoV2-1.1-S: 1 x 10^10 IU ± 0.5 Log: Healthy participants received VXA-CoV2-1.1-S at a dose of 1 x 10^10 IU ± 0.5 log as an oral tablet on Day 1 and Day 29 of the 57-day active study period.
- Active Study Period: VXA-CoV2-1.1-S: 1 x 10^11 IU ± 0.5 Log: Healthy participants received VXA-CoV2-1.1-S at a dose of 1 x 10^11 IU ± 0.5 log as an oral tablet on Day 1 and Day 29 of the 57-day active study period.
- Safety Follow-up Period: VXA-CoV2-1.1-S: 1 x 10^10 IU ± 0.5 Log: Healthy participants who received VXA-CoV2-1.1-S at a dose of 1 x 10^10 IU ± 0.5 log and entered the safety follow-up period until Month 13.
- Safety Follow-up Period: VXA-CoV2-1.1-S: 1 x 10^11 IU ± 0.5 Log: Healthy participants who received VXA-CoV2-1.1-S at a dose of 1 x 10^11 IU ± 0.5 log and entered the safety follow-up period until Month 13.
Arm/Group | Active Study Period: VXA-CoV2-1.1-S: 1 x 10^10 IU ± 0.5 Log | Active Study Period: VXA-CoV2-1.1-S: 1 x 10^11 IU ± 0.5 Log | Safety Follow-up Period: VXA-CoV2-1.1-S: 1 x 10^10 IU ± 0.5 Log | Safety Follow-up Period: VXA-CoV2-1.1-S: 1 x 10^11 IU ± 0.5 Log
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/21 | 1/44 | 0/21
Serious Adverse Events (participants affected / at risk) | 1/45 | 0/21 | 3/44 | 0/21
Other Adverse Events (participants affected / at risk) | 25/45 | 14/21 | 1/44 | 3/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active Study Period: VXA-CoV2-1.1-S: 1 x 10^10 IU ± 0.5 Log (N=45) | Active Study Period: VXA-CoV2-1.1-S: 1 x 10^11 IU ± 0.5 Log (N=21) | Safety Follow-up Period: VXA-CoV2-1.1-S: 1 x 10^10 IU ± 0.5 Log (N=44) | Safety Follow-up Period: VXA-CoV2-1.1-S: 1 x 10^11 IU ± 0.5 Log (N=21)
Hospitalization (Surgical and medical procedures) | 1 | 0 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Active Study Period: VXA-CoV2-1.1-S: 1 x 10^10 IU ± 0.5 Log (N=45) | Active Study Period: VXA-CoV2-1.1-S: 1 x 10^11 IU ± 0.5 Log (N=21) | Safety Follow-up Period: VXA-CoV2-1.1-S: 1 x 10^10 IU ± 0.5 Log (N=44) | Safety Follow-up Period: VXA-CoV2-1.1-S: 1 x 10^11 IU ± 0.5 Log (N=21)
COVID-19 (Infections and infestations) | 3 | 1 | 1 | 1
Amylase increased (Investigations) | 0 | 2 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 0 | 0
Thirst (General disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 11 | 5 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 4 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 4 | 3 | 0 | 0
Nausea (Gastrointestinal disorders) | 4 | 3 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 6 | 2 | 0 | 0
Malaise (General disorders) | 9 | 6 | 0 | 0
Fatigue (General disorders) | 7 | 5 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Vaxart decided not to conduct Part 2 of this study, so results for Part 2 were not included in this summary.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-04): https://cdn.clinicaltrials.gov/large-docs/33/NCT05067933/Prot_SAP_000.pdf